CLINICAL TRIAL: NCT02105064
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) as an add-on Treatment for Resistant Obsessive-compulsive Symptoms in Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10-0426
Record Dates: First submitted 2013-09-16; First posted 2014-04-07 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Schizophrenia; Obsessive-Compulsive Symptoms
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active rTMS (Active Comparator): rTMS over Supplementary Motor Area, 1hz, no pauses, 20 minutes per sessions. Total: 20 sessions.
  Interventions: Device: Active rTMS
- Sham (Sham Comparator): Sham stimulation, 20 minutes per session, total 20 sessions
  Interventions: Device: SHAM rTMS

INTERVENTIONS:
Device: Active rTMS — rTMS over supplementary motor area, 1hz, no pauses, 20 minutes/sessions, 5 sessions/week, 4 weeks. Total 20 sessions.
  Arms: Active rTMS
Device: SHAM rTMS — Sham rTMS, without brain stimulation
  Arms: Sham

SUMMARY:
This is a study to evaluate the efficacy of rTMS for relief of obsessive-compulsive symptoms in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Schizophrenia (DSM-IV-TR)
* YBOCS ≥ 16

Exclusion Criteria:

* Mental Retardation
* Substance abuse
* Any contraindication to rTMS

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-07; Primary Completion 2014-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change of Obsessive Compulsive symptoms (using Yale-Brown Obsessive Compulsive Scale - Y-BOCS) | Baseline, after 20 rTMS sessions (an expected average of 4 weeks), and 4 weeks after end of treatment

SECONDARY OUTCOMES:
Change of Psychotic Symptoms (using Brief Psychiatric Rating Scale - BPRS) | Baseline, after 20 rTMS sessions (an expected average of 4 weeks), and 4 weeks after end of treatment
Change of Brain-Derived Neurotrophic Factor (BDNF) | Baseline, after 20 rTMS sessions (an expected average of 4 weeks), and 4 weeks after end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided